CLINICAL TRIAL: NCT00814463
Title: Phase II Single-arm Study of Post-operative Stereotactic Radiosurgery for Brain Metastases.
Brief Title: Stereotactic Radiosurgery After Surgery in Treating Patients With Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early analysis indicated SRS not as beneficial post-op as pre-op
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00004373; DUMC-PRO00004373 (Other: DUHS IRB); CDR0000630239
Record Dates: First submitted 2008-12-23; First posted 2008-12-24 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: tumors metastatic to brain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms | interventions — Mental Status and Dementia Tests; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Post-operative SRS (Active Comparator): All patients will undergo SRS with the planned target volume (PTV) defined as the resection cavity plus a 3-mm margin after surgical resection of a single brain metastasis. Dose will be prescribed to the maximum isodose line completely encompassing the PTV using the guidelines established in RTOG 9005. All patients will be evaluated for neurocognitive function via Mini-Mental State Examination (MMSE), Quality of Life (QOL) via FACT-Br, and for local recurrence via MRI every 3 months over the course of the study.
  Interventions: Behavioral: MMSE; Behavioral: QOL via FACT-Br; Procedure: MRI; Radiation: Post-operative SRS

INTERVENTIONS:
Behavioral: MMSE — Neurocognitive function via MMSE done every 3 months for length of study.
  Other Names: Mini-Mental Status Exam
Behavioral: QOL via FACT-Br — Quality of Life via FACT-BR every 3 months for length of study.
  Other Names: Quality of Life; Functional Assessment of Cancer Therapy - Brain
Procedure: MRI — MRI done every 3 months for the length of the study.
  Other Names: Magnetic Resonance Imagine
Radiation: Post-operative SRS — Single fraction SRS is currently a viable treatment option of intracranial metastatic lesions.
  Other Names: SRS

SUMMARY:
RATIONALE: Stereotactic radiosurgery may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Giving stereotactic radiosurgery after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase II trial is studying how well stereotactic radiosurgery works in treating patients with brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To estimate the rate of recurrence at the surgical site in patients with brain metastases treated with adjuvant stereotactic radiosurgery (SRS) compared with historical data documenting recurrence at the surgical site after surgery and whole brain radiotherapy (WBRT).

Secondary

* To estimate the rate of salvage WBRT, SRS, or surgery in patients treated with adjuvant SRS alone.
* To estimate the rate of new brain metastases outside of the adjuvant SRS site.
* To estimate patient quality of life after adjuvant SRS alone.
* To assess the effect of surgical intervention and SRS on the preservation of neurocognitive functioning in these patients.
* To determine the clinical significance (if any) of locally recurrent brain metastases at the time of their occurrence (mass effect, cognitive functioning, and other symptoms) in these patients.
* To estimate the rate of death due to neurologic causes, defined as death attributable to the progression of neurological disease.
* To estimate the overall survival of these patients.

OUTLINE: Patients undergo stereotactic radiosurgery over 30-90 minutes.

Quality of life and neurocognitive function are assessed periodically.

After completion of study therapy, patients are followed every 3 months for 1 year and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years of age.
2. Gross total resection (as verified by the lack of any enhancement in the resection cavity on post-operative MRI) of single brain metastasis confirmed by histology. Patients with up to 4 metastases are eligible if the largest mass is amenable to surgical resection and all non-resected masses are amenable to SRS.
3. Patient must be Radiation Therapy Oncology Group (RTOG) recursive partitioning analysis (RPA) Class 1 or 2.
4. Life expectancy of at least 3 months.

Exclusion Criteria:

1. Radiographic or cytologic evidence of leptomeningeal disease.
2. Patient with incomplete or partial resection.
3. Primary lesion with radiosensitive histology (i.e., small cell carcinoma, germ-cell tumors, lymphoma, leukemia, and multiple myeloma).
4. Patients with a resection cavity > 4 cm in maximal extent in any plane on contrasted MRI scan.
5. Lesion located in anatomic regions which are not amenable to SRS including the brain stem and optic apparatus.
6. Pregnant or need to breast feed during the study period.
7. Uncontrolled intercurrent illness including, but not limited to symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness.
8. Brain surgery other than for resection of metastasis.
9. Previous brain radiotherapy.
10. Contraindication to SRS, WBRT, or MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John H. Sampson, MD, PhD, Principal Investigator — Duke University; Hamidreza Aliabadi, MD, Principal Investigator — Duke University; John P. Kirkpatrick, MD, Principal Investigator — Duke University; James E. Herndon, PhD, Principal Investigator — Duke University
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Duke Comprehensive Cancer Center from 6/12/2008 - 6/5/2009.
Groups:
- Post-operative SRS: All patients will undergo SRS with the planned target volume (PTV) defined as the resection cavity plus a 3-mm margin after surgical resection of a single brain metastasis. Dose will be prescribed to the maximum isodose line completely encompassing the PTV using the guidelines established in RTOG 9005. All patients will be evaluated for neurocognitive function via Mini-Mental State Examination (MMSE), Quality of Life (QOL) via FACT-Br, and for local recurrence via MRI every 3 months over the course of the study.
  QOL via FACT-Br : Quality of Life via FACT-BR every 3 months for length of study.
  Post-operative SRS : Single fraction SRS is currently a viable treatment option of intracranial metastatic lesions.
  MMSE : Neurocognitive function via MMSE done every 3 months for length of study.
  MRI : MRI done every 3 months for the length of the study.
Period: Overall Study
Arm/Group | Post-operative SRS
Started | 1
Completed | 0
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Post-operative SRS
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Rate at the Surgical Site as Measured by MRI
Description: The number of months for local recurrence via MRI
Time Frame: 12 months
Measure: Number; unit: Months
Arm/Group | Post-operative SRS
Number analyzed (Participants) | 1
Months | 3.5

2. Secondary Outcome: Rate of Salvage Whole-brain Radiotherapy, Stereotactic Radiosurgery (SRS), or Surgery
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Post-operative SRS
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Rate of New Brain Metastases Outside of the Adjuvant SRS Site
Time Frame: 12 months
Population: Data not collected due to subject withdrawal.
Arm/Group | Post-operative SRS
Number analyzed (Participants) | 0

4. Secondary Outcome: Quality of Life as Measured by the FACT-Br Subscales
Time Frame: Every 3 months for 12 months
Population: Data not collected due to subject withdrawal.
Arm/Group | Post-operative SRS
Number analyzed (Participants) | 0

5. Secondary Outcome: Preservation of Neurocognitive Function as Measured by the Mini-Mental State Exam
Time Frame: Every 3 months for 12 months.
Population: Data not collected due to subject withdrawal.
Arm/Group | Post-operative SRS
Number analyzed (Participants) | 0

6. Secondary Outcome: Clinical Significance (if Any) of Locally Recurrent Brain Metastasis at the Time of Their Occurrence (Mass Effect, Cognitive Functioning, and Other Symptoms)
Time Frame: 12 months
Population: Data not collected due to subject withdrawal.
Arm/Group | Post-operative SRS
Number analyzed (Participants) | 0

7. Secondary Outcome: Rate of Death Due to Neurologic Causes
Time Frame: 12 months
Population: Data not collected due to subject withdrawal.
Arm/Group | Post-operative SRS
Number analyzed (Participants) | 0

8. Secondary Outcome: Overall Survival
Time Frame: 12 months
Population: Data not collected due to subject withdrawal.
Arm/Group | Post-operative SRS
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Post-operative SRS
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes